CLINICAL TRIAL: NCT04877106
Title: Bioequivalence of Sitagliptin Phosphate/Metformin Hydrochloride Tablets in Healthy Chinese Subjects: A Single-dose and Two-period Crossover Study
Brief Title: Bioequivalence of Sitagliptin Phosphate/Metformin Hydrochloride Tablets in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DBH061L012017
Record Dates: First submitted 2021-04-26; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin Phosphate/metformin Hydrochloride Tablets (JANUMET®) (Active Comparator): JANUMET®, 50mg/850mg, batch no. M047893, manufactured by MSD Pharma (Singapore) Pte.Ltd
  Interventions: Drug: Sitagliptin Phosphate/metformin Hydrochloride Tablets(JANUMET®,50mg/850mg)
- Sitagliptin Phosphate/metformin Hydrochloride Tablets (Experimental): 50mg/850mg, batch no. 161006, manufactured by Tonghua Dongbao Pharmaceutical Co., Ltd.
  Interventions: Drug: Sitagliptin Phosphate/metformin Hydrochloride Tablets (50mg/850mg)

INTERVENTIONS:
Drug: Sitagliptin Phosphate/metformin Hydrochloride Tablets(JANUMET®,50mg/850mg) — The subjects randomly received single oral administration of Sitagliptin Phosphate/metformin Hydrochloride Tablets (JANUMET®, 50mg/850mg)
  Arms: Sitagliptin Phosphate/metformin Hydrochloride Tablets (JANUMET®)
Drug: Sitagliptin Phosphate/metformin Hydrochloride Tablets (50mg/850mg) — The subjects randomly received single oral administration of Sitagliptin Phosphate/metformin Hydrochloride Tablets (50mg/850mg)
  Arms: Sitagliptin Phosphate/metformin Hydrochloride Tablets

SUMMARY:
An open-label, randomized, single-dose, two-period, two-group, crossover study was conducted in 48 healthy Chinese volunteers under fasted or fed conditions (24 volunteers for each condition) to assess the bioequivalence between two formulations of Sitagliptin Phosphate/metformin Hydrochloride Tablets.

DETAILED DESCRIPTION:
The single-dose randomized, open-label, two-period crossover study was executed in the Phase I Clinical Research Center of the Affiliated Hospital of Qingdao University. This study was conducted to assess the bioequivalence of Sitagliptin Phosphate/metformin Hydrochloride Tablets in healthy Chinese subjects and estimate the pharmacokinetics profiles of Sitagliptin Phosphate/metformin Hydrochloride Tablets. An open-label, randomized, single-dose, two-period, crossover study was conducted in 48 healthy Chinese volunteers under fasted or fed conditions (24 subjects for each condition) to assess the bioequivalence between two formulations of Sitagliptin Phosphate/metformin Hydrochloride Tablets. Blood samples were collected at specified time intervals, and the plasma concentrations of sitagliptin and metformin were determined by a validated liquid chromatography mass spectrum/ mass spectrum method. Pharmacokinetic and bioavailability parameters were estimated via non-compartmental methods. Adverse events were also recorded. If the 90% confidence intervals of the ratios of geometrical mean of test and reference formulations for Cmax, AUC0-t and AUC0-∞ are all within the predefined bioequivalence criteria range of 80%-125% for sitagliptin and metformin, the two formulations can be considered bioequivalent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged between 18 and 45 years old (including the critical value).
* The body mass index is in the range of 19-28 kg/m2 (including the critical value). The weight of male is not less than 50 kg, and that of female is not less than 45 kg (including the critical value).
* Subjects who had not any medical history of cardiovascular, digestive, respiratory, nervous or hepatic/renal impairment. The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: physical examination, 12-lead ECG, vital sign measurements, and laboratory safety tests.
* The subjects have no family planning within 6 months and could select contraceptive method.
* Before the study, all subjects have been informed of the study's purpose, protocol, benefits, and risks, and signed the informed consent voluntarily.
* The subjects could complete the study according to the protocol.

Exclusion Criteria:

* Being allergy to the study medications, smoking, alcohol abuse.
* Participation in another clinical trial within 3 months.
* Any history of hypersensitivity, needlesickness or idiosyncratic reactions to any food or drug;
* Any use of other prescription drugs (including contraceptive) 14 days prior to medication for this study;
* Any use of prescription or over-the-counter drugs, functional vitamin, herbal/ alcohol products, grapefruit-containing or caffeine/xanthine-rich food and beverages 48 h prior to medication for this study; dysphagia or having special dietary requirements;
* occurring acute disease in the screening period or before the medication lactating or pregnant women;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-04-07 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The ratios of geometrical mean | 80 days
  The two preparations were considered bioequivalent if the 90% CIs of the ratios of the primary pharmacokinetics parameters were within the predefined acceptance range of 80%-125%.

SECONDARY OUTCOMES:
The occurrence rate of adverse events | 80 days
  Adverse events were recorded to evaluate the safety of the studied drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Doctor Cao, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shanndong, China

IPD SHARING:
Plan to Share IPD: No